CLINICAL TRIAL: NCT05350982
Title: A Prospective Feasibility Study of a Novel Salivary Collection Technique for the Measurement of Salivary Cortisol and Cortisone in Neonates, Infants and Toddlers
Brief Title: Neonatal, Infant and Toddler Salivary Study (NITS Study)
Acronym: NITS
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2596
Record Dates: First submitted 2021-11-25; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Adrenal Insufficiency
Keywords: Salivary collection; Salivary cortisol; Salivary cortisone
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital Arm: Participants will be recruited to use the SalivaBio +/- SaliPac in a hospital setting. They will be provided with collecting instructions and will be guided by a member of the research team.
  Interventions: Device: SalivaBio +/- SaliPac
- Stimulated Home Arm: 10 participants will be randomly selected by a random number generator. This arm will also be conducted in the Hospital, and the collection using a SalivaBio +/- SaliPac will still be observed by a member of the research team. These participants will receive the same information as those in the Hospital Arm, but will receive minimal input. This is to establish whether the collection instructions provided would be suitable to use in the home environment.
  Interventions: Device: SalivaBio +/- SaliPac

INTERVENTIONS:
Device: SalivaBio +/- SaliPac — Sterile collection swab (SalivaBio), Modified dummy (SaliPac)

SUMMARY:
Currently, the only way to analyse glucocorticoids for the screening or diagnosis of AI in young children is via plasma obtained by invasive capillary or venous blood sampling. Thus, there is an unmet need for a safe and simple salivary collection technique for use in children under the age of six years. The development of the SalivaBio offers potential for salivary collection, which is safe, easy and less-invasive than current practice. The SaliPac has been developed to offer a more tolerable and pleasant way of sampling saliva using a SalivaBio in very young children which the investigators envisage being used by parents/carers at home to sample and then post to the hospital for GC analysis.

DETAILED DESCRIPTION:
The adrenal glands sit above the kidneys and are part of the body's endocrine system. They produce a number of different steroid hormones; those involved in metabolism (glucocorticoids, principally cortisol and its more inactive form, cortisone), salt and water balance (aldosterone) and sex steroids (oestrogen and testosterone). Measurement of steroids, in particular glucocorticoids, in saliva rather than blood samples, is gaining popularity as it offers a non-invasive collection technique, enabling sampling in outpatients, the community or the home environment, and therefore an improved patient experience.

Adrenal insufficiency (AI) describes the inability of the body to produce adequate levels of the vital stress hormone, cortisol. It is associated with considerable mortality and morbidity. There are numerous causes, both in adults and children. The commonest cause in children is AI secondary to steroid medication prescribed for inflammatory conditions such as arthritis and asthma. AI is usually permanent but, especially in those patients taking steroid medication, it may not be, and repeated testing may be required. Testing for AI requires measurement of cortisol. Cortisol levels change during the day (highest soon after waking) and increase in response to stress. There is a lack of data on what constitutes a normal cortisol level under different conditions in children, especially babies and very young children. The investigators would like to use salivary glucocorticoid sampling to study normal responses in children, in order to be able to better define what is abnormal, to ensure appropriate and safe management of children at risk of AI in the future. The current salivary collection techniques (SCT) require active patient participation, present a potential choking hazard, and are therefore unsuitable for very young children. The investigators have been working on a SCT suitable for neonates, infants, and toddlers. Our novel SCT uses a salivary steroid swab encased in a pacifier/dummy (SaliPac) and will enable study of normal adrenal gland function at different ages and under different conditions and disease states from which the investigators will construct normal reference ranges. The final step in the validation of the novel SCT is this patient study where usability, patient tolerability and carer acceptability will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending Sheffield Children's Hospital Emergency Department, outpatients or a current inpatient
* Patients attending the hospital for any reason but well enough to participate in the study (determined by the clinical care team)
* Siblings of patients if appropriate
* Individuals of any sex
* Aged 5 years or under
* Informed consent from parent(s)/carer(s)

Exclusion Criteria:

* Aged 6 years or above
* Mouth pathologies e.g., ulcers, infection, abscesses, injury or pain

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 5 and under
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
To determine whether the SalivaBio ± SaliPac can be used to collect 1mL (optimal volume) of saliva from children aged five years and under in two minutes or under. | 2 minutes
  Salivary volume will be quantified by measuring change in mass of swab at start of collection compared to the end

SECONDARY OUTCOMES:
To assess whether the SalivaBio ± SaliPac supports collection of 0.2ml saliva (minimum volume required for analysis of salivary GC) in two minutes or under. | 2 minutes
  Salivary volume will be quantified by measuring change in mass of swab at start of collection compared to the end
To determine the acceptability of the SalivaBio ± SaliPac in participants (neonates, infants and toddlers) through parental opinion using a parental questionnaire ranked from 1-10 with 10 being the most acceptable to the parent | Within 10 minutes of sample collection
  Assessed through the use of parent/carer questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom

REFERENCES:
- [Derived] Tonge JJ, Keevil BG, Craig JN, Whitaker MJ, Ross RJ, Elder CJ. Salivary Steroid Collection in Children Under Conditions Replicating Home Sampling. J Clin Endocrinol Metab. 2022 Nov 23;107(11):3128-3136. doi: 10.1210/clinem/dgac419. PMID 35961299